CLINICAL TRIAL: NCT01864486
Title: Restoring Vision With the Intelligent Retinal Implant System (IRIS V1)in Patients With Retinal Dystrophy (Title in France: Compensation of Vision With the Intelligent Retinal Implant System (IRIS V1) in Patients With Retinal Dystrophy)
Brief Title: Restoring Vision With the Intelligent Retinal Implant System (IRIS V1)in Patients With Retinal Dystrophy
Acronym: IRIS-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Science Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP4M
Record Dates: First submitted 2013-05-15; First posted 2013-05-29 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Retinitis Pigmentosa; Cone Rod Dystrophy; Choroideremia
MeSH Terms: conditions — Retinitis Pigmentosa; Cone-Rod Dystrophies; Choroideremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intelligent Retinal Implant System (Experimental)
  Interventions: Device: Intelligent Retinal Implant System

INTERVENTIONS:
Device: Intelligent Retinal Implant System

SUMMARY:
This study evaluates the safety and effectiveness of the Intelligent Retinal Implants System (IRIS V1)

ELIGIBILITY:
Inclusion Criteria:

* Is 25 years or older at the date of enrolment
* Has a confirmed diagnosis of retinitis pigmentosa, choroideremia or cone-rod dystrophy
* Has a visual acuity of logMAR 2.3 or worse in both the eyes as determined by a Square Grating scale.
* Has functional ganglion cells and optic nerve activity
* Has a memory of former useful form vision
* Understands and accepts the obligation to present for all schedule follow-up visits.
* Has AP eye dimensions that are appropriate with the dimensions of the implant(In Germany: Has an AP eye dimension between 20.5 and 25 mm)
* Has head dimensions that are appropriate for visual Interface.

Exclusion Criteria:

* Has a history of severe glaucoma, uveitis, optic neuropathy or any confirmed damage to the optic nerve and/or visual cortex,
* Has any disease (other than study allowed diseases) or condition that affects retinal function of the study eye (e.g., central retinal artery/vein occlusion, end-stage diabetic retinopathy, current or prior retinal detachment, infectious or inflammatory retinal disease, etc.),
* Has any disease or condition that prevents adequate visualization of the retina of the study eye including, but not limited to, corneal degeneration that cannot be resolved prior to implantation,
* Has any disease or condition of the anterior segment of the study eye that prevents adequate physical examination (e.g., ocular trauma, etc.),
* Has severe nystagmus,
* Has any ocular condition that leads him or her to eye rubbing,
* Has any disease or condition that precludes the understanding or communication of the informed consent, study requirements or test protocols (e.g., deafness , multiple sclerosis, amyotrophc lateral sclerosis, neuritis, etc),
* Has a history of epileptic seizure,
* Has a history of chronic or recurrent infection or inflammation that would preclude participation in the study,
* Has a known sensitivity to the contact materials of the implant,
* Presents with hypotony in the study eye,
* Presents with hypertony in the study eye,
* Is pregnant or lactating,
* Has another active implanted device (e.g. cochlear implant) or any form of metallic implant in the head (other than dental work) that may interfere with the device function,
* Has a diagnosis requiring an active implant (e.g., cardiac pacemaker, vagus nerve implant, etc.),
* Has active cancer or a history of intraocular, optic nerve or brain cancer and metastasis,
* Is an immune-suppressed subject (e.g., due to HIV positive diagnosis, etc.),
* Is carrier of multi-resistant germs,
* Requires the use of any of the following medications:

  * Antimetabolites,
  * Thrombocyte aggregation reducing therapies (10 days prior until 3 days after surgery),
  * Oral anticoagulants (5 days before until 3 days after surgery),
* Is participating in another investigational drug or device study that may interfere with the proposed treatment or the ensuring follow-up schedule, (in Germany: Is participating in another investigational drug or device study)
* Has any health concern that makes general anaesthesia inadvisable, (in Germany: Patients with an ASA-Score of 3 or higher are excluded from the study)
* Is likely requiring MRI scans subsequent to implantation and prior to explantation,
* Is likely requiring therapeutic ultrasound subsequent to implantation and prior to explantation of the Retinal Implant

In Germany: - Patients with recurrent or chronic inflammations or infections are excluded from the study. Specifically patients with the following disorders are excluded:

* Common inflammation - severe chronic and consuming diseases that frequently associated with infection (e.g. Crohn disease, Whipple's disease)
* Chronic inflammation of the skin in the area of the eye (e.g. dermatitis, rosacea, infection of the skin, herpes zoster)
* Chronic inflammation in the area of the eye (e.g. herpes of cornea and/or conjunctiva, recurrent blepharoconjunctivitis, horedolum, chalazion) In Germany: - Has a severe psychological disorder. When in any doubt, an expert assessment needs to be arranged to clarify whether the patient's psychological health is suitable for the trial.

In Germany: - Has severe renal, cardiac, hepatic etc. organ diseases

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-10-13 (Actual); Study Completion 2017-10-13 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events as a Measure of Safety and Tolerability | Up to 18 month after implantation
  All subjects undergo ophthalmological examinations in predefined intervals after implantation. Ophthalmological examinations include funduscopy, slit lamp examination and OCT. All adverse events are recorded and analysed.

SECONDARY OUTCOMES:
Probable benefit | Up to 18 months after implantation
  A series of vision test including grating visual acuity, light localization and contrast sensitivity is performed before and after implantation of the device.

CONTACTS AND LOCATIONS:
Locations (5):
- Medical University of Graz, Graz, Austria
- France (2):
  - Clinique Ophtalmologique du CHU de Nantes, Nantes
  - Hopital des Quinze Vingts/Fondation Ophtalmologique A. De Rothschild, Paris
- Germany (2):
  - Dept. of Ophthalmology, University of Bonn, Bonn
  - Klinik und Poliklinik für Augenheilkunde Hamburg-Eppendorf, Hamburg